CLINICAL TRIAL: NCT02443844
Title: Comparison of Medical and Surgical Treatments of Benign Prostate Hyperplasia in Patients Who Have Low Grade Non Muscle Invasive Bladder Cancer for Tumour Recurrence and Progression
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Nihat Karakoyunlu, MD, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16.02.2015 20/03
Record Dates: First submitted 2015-04-28; First posted 2015-05-14 (Estimated); Last update posted 2015-05-14 (Estimated); Status verified 2015-05

CONDITIONS: Bladder Cancer
Keywords: BPH; bladder cancer; treatment; recurrence; progression
MeSH Terms: conditions — Urinary Bladder Neoplasms; Recurrence; Disease Progression | interventions — Tamsulosin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- First group (Active Comparator): Patients taken tamsulosin for benign prostate hyperplasia who have non muscle invasive bladder cancer
  Interventions: Drug: Tamsulosin
- Second Group (Active Comparator): Patients taken transurethral resection prostatectomy for benign prostate hyperplasia who have non muscle invasive bladder cancer
  Interventions: Procedure: Transurethral Resection

INTERVENTIONS:
Procedure: Transurethral Resection — Endoscopic treatment of bladder cancer
  Arms: Second Group
Drug: Tamsulosin — Medical treatment for benign prostate hyperplasia
  Other Names: alfa blocker treatment
  Arms: First group

SUMMARY:
The purpose of this study is to compare medical and surgical treatments of benign prostate hyperplasia in patients who have non muscle invasive bladder cancer for tumour recurrence and progression.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have non muscle invasive bladder cancer male patients patients between 40-80 years old

Exclusion Criteria:

* Patients who have previous prostate surgery Patients who have muscle invasive bladder cancer

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-02; Primary Completion 2018-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Recurrence | 3 years
  Bladder cancer recurrence rate

SECONDARY OUTCOMES:
Progression | 3 years
  Bladder cancer progression rate

CONTACTS AND LOCATIONS:
Overall Officials: Nihat Karakoyunlu, MD, Principal Investigator — Dıskapı TRH
Locations (1):
- Turkish Ministry of Health Dıskapı Yıldırım Beyazıt Training and Research Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Result] Li S, Zeng XT, Ruan XL, Wang XH, Guo Y, Yang ZH. Simultaneous transurethral resection of bladder cancer and prostate may reduce recurrence rates: A systematic review and meta-analysis. Exp Ther Med. 2012 Oct;4(4):685-692. doi: 10.3892/etm.2012.660. Epub 2012 Aug 9. PMID 23170127